CLINICAL TRIAL: NCT00405847
Title: A Pilot Study of Effect of Dexmedetomidine on Sleep and Inflammation in Critically Ill Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Arizona (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: HSC #06-107
Record Dates: First submitted 2006-11-29; First posted 2006-11-30 (Estimated); Last update posted 2016-10-27 (Estimated); Status verified 2016-10

CONDITIONS: Sleep; Critical Illness
Keywords: Sleep; Critical illness; Cytokine
MeSH Terms: conditions — Critical Illness | interventions — Dexmedetomidine

INTERVENTIONS:
Drug: Dexmedetomidine

SUMMARY:
The purpose of this study is to assess the short-term effect of sympatholysis on sleep quality and inflammation in critically ill patients.

DETAILED DESCRIPTION:
Over 1 million patients receive mechanical ventilation every year in the United States. In mechanically ventilated patients, despite sedative infusions, sleep is severely disrupted. Sleep disruption, in turn, can lead to activation of sympathetic nervous system and elevated inflammatory cytokines. Both sympathetic hyperactivity and elevated cytokines have been associated with delirium, which, in turn, is associated with increased mortality and higher healthcare costs. Currently, however, there is very little understanding of the inter-relationship between critical illness, sleep, and neuropsychological well-being. The purpose of this study is to collect preliminary data on the short-term effects of sedation with and without sympatholysis on sleep and inflammation in critically ill patients receiving mechanical ventilation. This pilot study will be accomplished by performing sleep studies and circulating cytokine measurements in critically ill patients randomized to receive two different sedation strategies: Dexmedetomidine versus Midazolam and Fentanyl. The ultimate goal of this program of research is to identify sedation practices that are least associated with adverse short- and long-term consequences, and thereby ultimately help improve sleep quality and quality of life in patients surviving critical illness.

ELIGIBILITY:
Inclusion Criteria:

* Patients requiring mechanical ventilation with a diagnosis of

  * Acute Respiratory Distress Syndrome
  * Cardiogenic Pulmonary Edema
  * Pneumonia
  * Chronic obstructive pulmonary disease

Exclusion Criteria:

* Patients who are considered too unstable to undergo this investigation by their primary physician
* Comatose patients, or patients with severe debilitating neurological disease
* Renal insufficiency (Sr. Creatinine > 2 mg/dL)
* Heart block (second or third degree heart block) or sinus bradycardia (heart rate < 60 beats per minute)
* Pregnancy

Ages: 21 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2006-07; Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
Sleep disruption (Arousals, awakenings and sleep efficiency measured by polysomnography)
Circulating levels of Inflammatory cytokines (TNF-alpha, IL-1, IL-6, IL-10)

CONTACTS AND LOCATIONS:
Overall Officials: Sairam Parthasarathy, MD, Principal Investigator — SAVAHCS and University of Arizona
Locations (1):
- Southern Arizona VA Healthcare System, Tucson, Arizona, United States